CLINICAL TRIAL: NCT02798861
Title: Usefulness of Controlled Attenuation Parameter (CAP) for the Assessment of Liver Steatosis in Liver Donors
Brief Title: Controlled Attenuation Parameter (CAP) in Liver Allografts
Status: Completed | Type: Observational
Sponsor: Andres Duarte-Rojo (Other)
Responsible Party: Sponsor-Investigator, Andres Duarte-Rojo, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: 204560
Record Dates: First submitted 2016-06-02; First posted 2016-06-14 (Estimated); Results first posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Liver Transplant; Liver Steatosis; Liver Disease; Primary Non-function; Early Allograft Dysfunction
MeSH Terms: conditions — Fatty Liver; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CAP assessment: Controlled Attenuation Parameter with Fibroscan 402/530 before liver procurement and after liver transplantation to assess steatosis, and its association with clinical outcomes
  Interventions: Device: Fibroscan 402/530

INTERVENTIONS:
Device: Fibroscan 402/530 — Fibroscan 402/530 obtained before procurement in the donor and at 1 to 3 months post-transplant in the liver recipient.

SUMMARY:
The primary aim is to determine the accuracy of CAP in the quantification of liver steatosis using liver biopsies as reference. Secondarily, investigators will correlate transient elastography (TE) and CAP results, analyze possible associations between CAP/TE and post-liver transplant (LT) clinical outcomes, and evaluate the change in CAP after LT. The study aims to include as many donors as needed to achieve at least 120 transplanted liver allografts.

DETAILED DESCRIPTION:
This is a coordinated study utilizing 3 recruitment centers (University of Arkansas for Medical Sciences [UAMS], Stanford University, and Mayo Clinic) 2 liver pathology reading centers (University of Michigan and Mayo Clinic), and 1 coordinating center (University of Arkansas). The cohort study with a cross-sectional component for the primary aim has been completed (through independent Institutional Review Board [IRB] agreements) at UAMS, Stanford University, and the Mayo Clinic. The samples collected at the three recruitment centers will be sent to the biopsy center at the University of Michigan and Mayo Clinic for evaluation. The Liver Transplant Program at each of the 3 recruiting centers will identify study subjects during the process of liver allocation to their listed recipients. Criteria for recruitment are as follows:

Inclusion criteria - Liver Recipient

* Men and women, Age 18-years old to 80-years old inclusive Inclusion criteria - Liver Donor
* Valid TE with Fibroscan 530, defined as:

  * At least 10 valid measurements
  * Interquartile Range (IQR)/Median stiffness value <30% (only in cases with >7.1 kPa) Exclusion criteria - Liver Recipient
* Patient did not undergo liver transplantation Exclusion criteria - Liver Donor
* Donation after circulatory death (DCD)
* No liver biopsy obtained during organ procurement process

ELIGIBILITY:
Inclusion criteria - Liver Recipient

* Men and women, Age 18-years old to 80-years old inclusive

Inclusion criteria - Liver Donor

* Valid TE with Fibroscan 402/530, defined as:

  * At least 10 valid measurements
  * IQR/Median stiffness value <30% (only in cases with >7.1 kPa)

Exclusion criteria - Liver Recipient

* Patient did not undergo liver transplantation

Exclusion criteria - Liver Donor

* Donation after circulatory death (DCD)
* No liver biopsy obtained during organ procurement process

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Allograft procured and transplanted into recipients.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Duarte-Rojo, MD, Principal Investigator — University of Pittsburgh
Locations (3):
- United States (3):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Stanford University, Stanford, California
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Allografts: Livers assessed before procurement and after implantation.
Period: Overall Study
Arm/Group | Allografts
Started | 160
Completed | 137
Not Completed | 23
Not completed — Lost to Follow-up | 22
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | CAP Assessment
Number analyzed (Participants) | 160
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 116
  Race/Ethnicity: Black | 22
  Race/Ethnicity: Hispanic | 3
  Race/Ethnicity: Asian | 2
  Race/Ethnicity: Other | 3
  Race/Ethnicity: Unknown | 14
Region of Enrollment [Number; unit: participants]
  United States | 160
ALT [Median (Inter-Quartile Range); unit: IU/L] | 36 [21 to 90]
AST [Median (Inter-Quartile Range); unit: IU/L] | 83 [43 to 195]
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27 (6)
CAP [Median (Inter-Quartile Range); unit: dB/m] | 235 [188 to 274]
LSM [Median (Inter-Quartile Range); unit: kPa] | 7.25 [5.7 to 10.2]

OUTCOME MEASURES:

1. Primary Outcome: Controlled Attenuation Parameter (CAP) - Accuracy
Description: CAP accuracy in quantification of liver steatosis to be determined using liver biopsies as reference
Time Frame: Baseline (pre-procurement) to 6 months post liver transplant
Population: Here are considered the allografts that were transplanted and whose recipients consented to participate in study
Measure: Median (Inter-Quartile Range); unit: dB/m
Groups:
- CAP Assessment: Controlled Attenuation Parameter with Fibroscan 402/530 before liver procurement and after liver transplantation to assess steatosis, and its association with clinical outcomes
  Fibroscan 402/530: Fibroscan 402/530 obtained before procurement in the donor and at 1 to 6 months post-transplant in the liver recipient.
Arm/Group | CAP Assessment
Number analyzed (Participants) | 110
dB/m | 220 [176 to 262]

2. Secondary Outcome: LSM
Description: Liver stiffness measurement
Time Frame: Pretransplant to 6 months posttransplant
Population: Here are considered the allografts that were transplanted and whose recipients consented to participate in study
Measure: Median (Inter-Quartile Range); unit: kPa
Arm/Group | CAP Assessment
Number analyzed (Participants) | 110
kPa | 6 [4.7 to 8.7]

ADVERSE EVENTS:
Time Frame: No adverse event data were collected because the study was observational.
Description: No adverse event data were collected because the study was observational.
Arm/Group | CAP Assessment
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT02798861/Prot_SAP_000.pdf